CLINICAL TRIAL: NCT04221191
Title: Study on the Dimethyl Fumarate (DMF, Tecfidera®) Persistence of Remitting-relapsing Multiple Sclerosis (RR-MS) Patients Included in the French Patient Support Program (PSP) OroSEP
Brief Title: Dimethyl Fumarate (DMF, Tecfidera®) Persistence in RR-MS Patients Included in the French Patient Support Program OroSEP
Acronym: TEC-ADHERE
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: FRA-BGT-18-11469
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of Care (SoC) Group: SoC neurologists will include and follow-up all study participants who receive DMF according to their standard of care practice (non-coached participants).
  Interventions: Drug: Dimethyl Fumarate
- OroSEP PSP (OPSP) Group: OPSP neurologists will include and follow-up all study participants who receive DMF according to their standard of care practice and the OroSEP PSP (coached participants).
  Interventions: Drug: Dimethyl Fumarate; Other: PSP

INTERVENTIONS:
Drug: Dimethyl Fumarate — DMF as prescribed as standard of care.
  Other Names: Tecfidera®
Other: PSP — PSPs is to support patient care.
  Groups: OroSEP PSP (OPSP) Group

SUMMARY:
The primary objective is to compare oral dimethyl fumarate (DMF) persistence at six months in relapsing-remitting multiple sclerosis (RR-MS) participants initiating DMF with and without OroSEP patient support program (PSP), respectively.

The secondary objectives are: to compare oral DMF persistence at one month and three months in RR-MS participants initiating DMF with and without OroSEP PSP, respectively; To compare oral DMF adherence at six months in RR-MS participants initiating DMF with and without OroSEP PSP; To compare at three months and six months the reason of oral DMF discontinuation, in the two groups; To describe the percentage of participants with treatment-related adverse events globally and by class of adverse events, in the two groups of participants; To assess the evolution of participants' anxiety globally and to compare it at inclusion and at six months in participants with and without OroSEP PSP, respectively; To describe participants' satisfaction regarding oral DMF initiation and follow-up globally at six months and to compare it in patients with and without OroSEP PSP, respectively;

For OroSEP PSP group: To assess participants' satisfaction regarding their participation in OroSEP PSP at six months; To assess neurologists' satisfaction regarding their participation in OroSEP PSP, after the last participant last visit of center.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and giving oral informed consent regarding TEC-ADHERE study and authorization to use protected health information (PHI) in accordance with national and local participant privacy regulations;
* Diagnosis of RR-MS;
* Initiating oral DMF according to Summary of Product Characteristics (SmPC) at the inclusion visit;
* Expanded Disability Status Score (EDSS) under 6.

Key Exclusion Criteria:

* Participants with progressive form of Multiple Sclerosis (MS);
* With memory or psychiatric disorders preventing them to complete questionnaires in the study.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study population included participants with RR-MS treated with DMF in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Oral Dimethyl Fumarate (DMF) Persistence at 6 Months | 6 months
  Persistence is defined as the percentage of participant still being treated by oral DMF at 6 months, according to routine visit.

SECONDARY OUTCOMES:
Percentage of Participants with Oral Dimethyl Fumarate (DMF) Persistence at Both 1 Month and 3 Months | 1 month and 3 months
  Persistence is defined as the percentage of participants still being treated by oral DMF at both 1 month and 3 months, according to routine practice.
Percentage of Participant's with Adherence at 6 Months | 6 months
  Participant's adherence is assessed through the validated Girerd questionnaire. This is a 6-item self-questionnaire completed by participants with a scale of 0 for "Yes" and 1 for "No" for each question. Points for each question are summed up to obtain a global score between 0 if all the questions are ticked with "Yes" (reflecting a bad adherence), and 6 if all questions are ticked "No" (reflecting a good adherence).
Percentage of Participants by Reason of Oral Dimethyl Fumarate (DMF) Discontinuation at 3 Months and 6 Months | 3 month and 6 months
  Discontinuation of DMF therapy is defined by the presence of any of the following criteria: definitive discontinuation declared by the physician during routine follow-up visit through electronic case report form (eCRF); a temporary stop declared by the physician during routine visit at 3 months, without DMF resumption declared at 6 months by the physician; a switch to another DMT declared by the physician during routine follow-up visit through eCRF.
Percentage of Participants with Adverse Events (AEs) | up to 6 months
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Percentage of Participants with Adverse Events (AEs) Related to Treatment | up to 6 months
Percentage of Participants with Adverse Events (AEs) Leading to Treatment Discontinuation | up to 6 months
Percentage of Participants with Adverse Events (AEs) of Interest | up to 6 months
  AEs of interest includes gastrointestinal disorders, flush, lymphopenia.
Participant's Anxiety at Inclusion and at 6 Months | 0 months and 6 months
  Participant's anxiety is assessed through the Generalized Anxiety Disorder - 7 (GAD-7) self-questionnaire. The GAD-7 is a questionnaire that is used primarily to detect possible generalized anxiety disorders, disorders of panic, social anxiety and post-traumatic stress disorder. It is more specifically a self-questionnaire (completed by the participant) consisting of 7 items rated from 0 to 3. The total score is obtained by adding the score obtained to each item (score ranging from 0 to 21). A total score greater than 7 is suggestive of a generalized anxiety disorder.
Participant's Satisfaction Regarding Dimethyl Fumarate (DMF) Treatment at 6 Months | 6 months
  Participant's satisfaction regarding DMF treatment is assessed through the validated Treatment Satisfaction Questionnaire for Medication (TSQM-9) score completed by the participant. The TSQM-9, a 9-items questionnaire, designed as a general measure of treatment satisfaction with medication. TSQM items are answered on 5- or 7-point Likert type scale and cover three domains, corresponding to distinct aspects related to the satisfaction of participants with their treatment (effectiveness, convenience and global satisfaction). A score can be obtained for each domain by summing the corresponding items transformed on a 0-100 scale. Higher value indicates more satisfaction, better perceived effectiveness, lower burden associated with better convenience.
Participant's Satisfaction Regarding their Participation in OroSEP Patient Support Program (PSP) | 6 month
  Participant's satisfaction is assessed at Month 6 using a questionnaire completed by the participant consisting of 3 questions. Questions 1 and 2 are assessed using a Likert scale (1-5) with scale range 1= Strongly disagree to 5= Strongly agree. Question 3 is assessed using the net promoter scale (1-7), where 1 indicates "not at all likely" and 7 indicates "extremely likely". Higher values indicate higher satisfaction.
Neurologists' Satisfaction Regarding their Participation in OroSEP Patient Support Program (PSP) | up to 6 months
  Neurologist's satisfaction is assessed after the last participant last visit of the site center using a 10-item questionnaire, completed by the physician. Question (Q) 1, Q3, Q4, Q6, Q7, Q8= is answered "Yes/No"; Q2= Lack of time, Lack of interest, Patient refused, Forget, No registration form available, Registration process too complicated / Other: specify; Q5= The availability of the call center, The monitoring of patient compliance, The coordination of biological assessments, Other: specify; Q9: 1 bad satisfaction, 10 good satisfaction and Q10 was an open answer.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (63):
- France (63):
  - Ch D'Agen, Agen
  - CH d'Aix-en-Provence, Aix-en-Provence
  - CHU Amiens, Amiens
  - CHU D'amiens, Amiens
  - Cabinet Medical, Angoulême
  - Cabinet Medical Neurolac, Annecy
  - CH Antibes, Antibes
  - Hopital Prive Antony, Antony
  - CH d'Arras, Arras
  - CH de Bastia, Bastia
  - Chic de Bayonne, Bayonne
  - Cabinet du Dr Imad Malkoun, Belfort
  - Cabinet des Drs Chanel-Soulier et Cheron, Biarritz
  - Hôpital Pellegrin / Service : Neurologie, Bordeaux
  - Polyclinique Bordeaux-Caudéran, Bordeaux
  - Ch de Carcassonne, Carcassonne
  - Cabinet des Drs Farhat et Samad, Châtellerault
  - Chde Cholet, Cholet
  - HIA Percy, Clamart
  - Pole de Sante Du Plateau, Clamart
  - Clinique Des Cedres, Cornebarrieu
  - Hopital Henri Mondor, Créteil
  - Ch General Dax, Dax
  - Cabinet du Dr Pierre Gras, Dijon
  - CHU Dijon, Dijon
  - Ch de Douai, Douai
  - CH Simone Veil d'Eaubonne, Eaubonne
  - Cabinet de Dr Lotfi Kort, Évreux
  - Polyclinique des Alpes du Sud, Gap
  - CHU Grenoble Alpes CS 10217, Grenoble
  - Cabinet médical, La Rochelle
  - Pôle Espace Santé 2, La Seyne-sur-Mer
  - Centre Hospitalier de Libourne, Libourne
  - Cabinet médical Montebello, Lille
  - Centre Hospitalier Intercommunal JURA-SUD, Lons-le-Saunier
  - Chi de Haute Saone, Lure
  - Cabinet Du Dr Neuschwander, Lyon
  - Hopital, Melun
  - CH de Montauban, Montauban
  - Centre Medical Odysseum, Montpellier
  - Hopital Gui de Chaulliac, Montpellier
  - Cabinet des Drs Lorenzi Pernot et Guilloton, Mornant
  - Clinique d'Occitanie, Muret
  - Chu Caremeau, Nîmes
  - CHU Carémeau, Nîmes
  - Hôpital de la Source, Orléans
  - Centre Cosem Miromesnil, Paris
  - Cabinet du Dr Radia Djebbari, Paris
  - Groupe Hospitalier Paris St Joseph, Paris
  - Cabinet Médical Monceau, Paris
  - Cabinet médical, Pau
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Chi de Cornouaille, Quimper
  - Cabinet des Drs Gugenheim et Esna, Rambouillet
  - Cabinet Du Dr Christophe Robin, Roanne
  - Hopital Victor Provo, Roubaix
  - CH de Soissons, Soissons
  - Cabinet du Dr Annick Gayou-Joyeux, Talence
  - HIA Sainte Anne, Toulon
  - Hopital Pierre-Paul Riquet, Toulouse
  - CHU Bretonneau, Tours
  - CH de Troyes, Troyes
  - CH de Valence, Valence

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Labauge P, Creange A, Moreau T, Nouvet-Gire J, Pedespan B, Heinzlef O, Texier N, Gros M, Marti C, Ruiz M, Martinez M, Castelnovo G. TEC-ADHERE: Real-World Persistence and Adherence on Dimethyl Fumarate in Patients with Relapsing-Remitting Multiple Sclerosis in the French OroSEP Patient-Support Program. Neurol Ther. 2025 Feb;14(1):177-192. doi: 10.1007/s40120-024-00674-x. Epub 2024 Nov 11. PMID 39527163